CLINICAL TRIAL: NCT07109544
Title: Effect of Breathing Exercises on Embryo Transfer Success Rates in In Vitro Fertilization Treatment: A Prospective Randomized Controlled Trial
Brief Title: Effect of Breathing Exercises on Embryo Transfer Outcomes
Acronym: BreathIVF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eurofertil IVF Health Center (Other)
Responsible Party: Principal Investigator, Elif Güler Ergin, Dr, Embryologist, Eurofertil IVF Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: eurofertil-breathing
Record Dates: First submitted 2025-07-18; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Pregnancy Outcomes
Keywords: Breathing exercises; IVF; Embryo transfer; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: As the possible effects of breathing exercises are planned to be analyzed, two groups are established. The groups are going to be formed by randomisation. While one group of patients will receive breathing exercises throughout their process , the control group patients will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy group (Experimental): The arm that the patients will receive breathing exercise therapy
  Interventions: Other: Breathing Therapy
- Control Arm (Other): The patients with standart care
  Interventions: Other: Breathing Therapy

INTERVENTIONS:
Other: Breathing Therapy — The patients in the control group will be receiving breathing therapy by a certificated clinical nurse

SUMMARY:
Breathing exercises are being used in many different clinical issues in the area of medicine. Also in gynecological practice, especially during labor, breathing exercises are encouraged by health professionals to aid the patients. These may have benefits of process of labor as it promises attenuating the anxiety and also relaxing the pelvic muscles. IVF, which may be one of most challenging times of couples, particularly women, is reported to be related with increased anxiety. Breathing exercises may potentially help women overcome anxiety before embryo transfer, a critical step in IVF. Being an easy and non-expensive approach, breathing exercises can be recommended in every IVF clinic. Thus, the investigators wanted to observe the effects of breathing exercises on embryo transfer results.

DETAILED DESCRIPTION:
The connection between breathing, especially abnormal breathing patterns, and emotions has always attracted attention and has been studied in various ways. There are publications reporting that this situation becomes even more evident when symptoms are associated with anxiety. Emotions are clearly expressed through breathing changes in rhythm, depth, location or regularity. It has been reported that the rhythm related to breathing is lost when there is a period of uncertainty for the person, especially in the near future. From this relationship, the possible positive effects of optimizing movements, breathing patterns and rhythms on emotional states can be expected. Breathing exercises and their effects have been investigated in many different patient groups in the field of medicine and their positive effects have been found.

This interest has also been observed in the field of obstetrics and gynecology. In a study published in 2023 examining the effects of breathing exercises on patients interned for birth, it was reported that breathing exercises increased the rate of normal birth and reduced the rate of caeserean section after labor, and also decreased the time spent for normal birth. Having a child is very important for couples. Therefore, not having a child is often observed as a distressing and worrying experience for couples. This situation can be expected to be even more pronounced, especially in couples who cannot achieve pregnancy after different treatments and trials and who reach the in vitro fertilization process.

There are also studies in the literature on the effect of the emotional state of couples, especially women, on the in vitro fertilization process . Different approaches have been put forward for the increased anxiety seen in these studies, and it has been shown that yoga and some other holistic medical practices can reduce the anxiety levels of women undergoing the in vitro fertilization process . However, to our knowledge, no study has drawn attention in which the possible benefits of breathing therapy have been examined in patients undergoing embryo transfer. The investigators aimed to investigate the effectiveness of breathing therapy, which is easy to apply and does not require any cost, in women who are potentially nervous or anxious due to embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* good quality blastocyst transfer

Exclusion Criteria:

* known psychiatric disorder
* history of recurrent implantation failure or pregnancy loss
* known genetik abnormalities
* known mullerian anomalies except for arcuate uterus
* PGT-a cycles

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only women having desire to achieve pregnancy who admitted to an IVF clinic
Enrollment: 100 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Pregnancy results after embryo transfer | 12 days after the embryo transfer
  Blood samples will be taken for beta-HCG test

CONTACTS AND LOCATIONS:
Overall Officials: Gerçek Aydın, Asst. Prof., Principal Investigator — Eurofertil IVF Health Center
Locations (1):
- Bursa Eurofertil IVF Center, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The names of patients will not be shared. The data of study can be shared upon request